CLINICAL TRIAL: NCT01592760
Title: Comparison of the Air-Q® Self-Pressurizing (SP) Intubating Laryngeal Airway With the Air-Q® Intubating Laryngeal Airway and I-gel for Airway Maintenance in Adults Under General Anesthesia
Brief Title: Air-Q® SP Versus Air-Q® and I-gel: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0805
Record Dates: First submitted 2012-05-02; First posted 2012-05-07 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-02

CONDITIONS: Laryngeal Masks
Keywords: air-Q SP; air-Q; i-gel; supraglottic airway device; laryngeal mask airway

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- air-Q SP (Experimental): air-Q Self-Pressurizing Intubating Laryngeal Airway, sizes 3.5 and 4.5 (Mercury Medical, Clearwater, FL, USA)
  Interventions: Device: air-Q SP
- air-Q (Active Comparator): air-Q Intubating Laryngeal Airway, sizes 3.5 and 4.5 (Mercury Medical, Clearwater, FL, USA)
  Interventions: Device: air-Q
- i-gel (Active Comparator): i-gel, sizes 3, 4, and 5 (Intersurgical Inc., Liverpool, NY, USA)
  Interventions: Device: i-gel

INTERVENTIONS:
Device: air-Q SP — air-Q SP placement for airway maintenance.
  Arms: air-Q SP
Device: air-Q — air-Q placement for airway maintenance.
  Arms: air-Q
Device: i-gel — i-gel placement for airway maintenance.
  Arms: i-gel

SUMMARY:
The air-Q Self-Pressurizing Intubating Laryngeal Airway (aILA SP) is a modification of the air-Q Intubating Laryngeal Airway (aILA). Besides the i-gel, it is the only breathing tube that sits above the vocal cords that does not require inflation of a cuff with air. The purpose of this study is to compare the ability of the aILA-SP to maintain patency of a patient's airway during general anesthesia with that of the aILA and i-gel devices. As a measure of this ability, we hypothesized that the airway sealing pressures will be equal between the aILA-SP and aILA, but superior when comparing the aILA-SP to the i-gel (i-gel will be lower).

DETAILED DESCRIPTION:
Laryngeal mask airways (LMAs) are a group of airway devices, alternatively referred to as supraglottic airways (SGAs), used in anesthesia that are positioned in the back of the throat (pharynx) above (supra) the glottis (windpipe opening) and the vocal cords. This is in contradistinction to a tracheal tube, which is an airway device that is placed through the vocal cords and extends to a position below the glottis (infraglottic) and resides in the trachea (windpipe). Since their first approval for use in the United States by the US Food and Drug Administration in the early 1990s, the application of SGAs has become more widespread. Initially, they were only used in anesthetized patients who were breathing on their own (i.e., spontaneously ventilating). This was, in large part, due to a relatively low airway seal pressure, the pressure with which the device seals against the throat, thereby, keeping the air pushed in by a breathing machine (ventilator) from getting into the stomach or leaking out around the device and out through the mouth - in either case, not going into the patient's lungs. The relatively low airway seal pressure (18 - 20 cmH2O) did not allow for the use of muscle relaxant (paralyzing) drugs and positive pressure ventilation. Successive generations of SGAs by a variety of manufacturers have overcome and continue to attempt to overcome limitations of earlier devices. In addition, accumulated clinical experience has made anesthesia providers more comfortable with their use. No SGA, however, is yet ideal, and incremental changes continue to appear to improve airway management and reduce airway morbidity (e.g., sore throat, jaw pain, etc.).

The air-Q® Intubating Laryngeal Airway (aILA, Mercury Medical, Clearwater, FL) is a newer, commercially-available, SGA designed for use as a primary airway and as an intubation conduit. It is available in polyvinyl chloride (PVC)-based, single use and silicone-based, reusable models. Information on its safety and effectiveness from a randomized, controlled trial in adults, undergoing general anesthesia, compared to that of the silicone-based, reusable aILA versus the LMA-Proseal™ (pLMA, North America, San Diego, CA), the current "gold standard" for SGA airway seal pressure, is available.

The air-Q® Self-Pressurizing (SP) Intubating Laryngeal Airway (aILA-SP, Mercury Medical, Clearwater, FL) is a commercially-available, modification of the silicone-based, reusable aILA. Its overall design is identical to the aILA, but incorporates a communication orifice between the air tube and cuff, which regulates airflow into and from the cuff during periods of positive pressure and spontaneous ventilation. As such, it incorporates a self-pressurizing cuff that does not require manual inflation. Such a cuff may be advantageous insofar as it dynamically adjusts its intra-cuff pressure and fit with the patient's pharyngeal and periglottic anatomy, which may lead to a reduction in airway morbidity, while still providing the high seal pressure afforded by the aILA design.

Lastly, the i-gel (Intersurgical Inc., Liverpool, NY) is a commercially-available SGA that uses a thermoplastic elastomer to create a non-inflating, anatomically-conforming, periglottic cuff. Studies have shown it to be an easily inserted, effective airway device with a lower incidence of sore throat and neck complaints. With exception to the aILA-SP, it is the only other commercially-available SGA that does not require cuff inflation.

To date, no reports are available on the clinical performance of the aILA-SP in relation to other SGAs. Thus, the primary purpose of this study is to compare the airway seal pressure (ASP) of the aILA-SP against the aILA and i-gel in adults undergoing general anesthesia. Airway seal pressure is the most common surrogate for ventilatory capacity used in SGA studies.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years;
* scheduled for an elective surgery or procedure; and
* general anesthesia with placement of a SGA planned.

Exclusion Criteria:

* < 18 years of age;
* non-English speaking;
* known or believed to be pregnant;
* prisoner;
* has impaired decision-making capacity;
* has symptomatic untreated gastroesophageal reflux;
* has had a prior esophagectomy;
* has a known or suspected hiatal hernia;
* has vomited within twenty-four hours of the surgery or procedure;
* has known oral pathology making a proper SGA fit unlikely; or
* has any condition for which the primary anesthesia care team deems intubation with a tracheal tube to be necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Galgon, MD, MS, Principal Investigator — Department of Anesthesiology, University of Wisconsin School of Medicine and Public Health
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable. There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Galgon RE, Schroeder KM, Han S, Andrei A, Joffe AM. The air-Q((R)) intubating laryngeal airway vs the LMA-ProSeal(TM) : a prospective, randomised trial of airway seal pressure. Anaesthesia. 2011 Dec;66(12):1093-100. doi: 10.1111/j.1365-2044.2011.06863.x. Epub 2011 Aug 22. PMID 21880031

RESULTS

PARTICIPANT FLOW:
Groups:
- Air-Q: Subjects randomized to receive air-Q for airway maintenance under general anesthesia.
- Air-Q SP: Subjects randomized to received an air-Q SP for airway maintenance under general anesthesia.
- I-gel: Subjects randomized to receive an I-gel for airway maintenance under general anesthesia.
Period: Perioperative to Discharge
Arm/Group | Air-Q | Air-Q SP | I-gel
Started | 90 | 90 | 45
Completed | 90 | 90 | 45
Not Completed | 0 | 0 | 0
Period: 24-hour Follow-Up
Arm/Group | Air-Q | Air-Q SP | I-gel
Started | 90 | 90 | 45
Completed | 86 | 87 | 43
Not Completed | 4 | 3 | 2
Not completed — Lost to Follow-up | 4 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Air-Q: air-Q Intubating Laryngeal Airway, sizes 3.5 and 4.5 (Mercury Medical, Clearwater, FL, USA)
  air-Q SP: air-Q SP placement for airway maintenance.
- Total: Total of all reporting groups
Arm/Group | Air-Q | Air-Q SP | I-gel | Total
Number analyzed (Participants) | 90 | 90 | 45 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14) | 45 (16) | 40 (15) | 43 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 41 | 15 | 88
  Male | 58 | 49 | 30 | 137
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28 (6) | 27 (5) | 27 (5) | 27 (5)
Mallampati Score [Number; unit: participants] — Mallampati Class is used to predict the ease of endotracheal intubation. Scores go from class 1 to class 4, where class 1 is the easiest intubation and class 4 is the most difficult. In order to measure Mallampati class, the standard approach to grading Mallampati class was used. Specifically, the investigator looked into the subject's oral opening facing the subject at a 90 degree angle and observed the appearance of the soft palate and extent of the uvula, while the subject fully extended the tongue from the oral cavity.
  participants
    Class 1 | 41 | 33 | 17 | 91
    Class 2 | 43 | 42 | 25 | 110
    Class 3 | 4 | 11 | 2 | 17
    Class 4 | 0 | 1 | 1 | 2
    Missing Data | 2 | 3 | 0 | 5
Device Size [Number; unit: participants]
  3 | 0 | 0 | 2 | 2
  3.5 | 32 | 42 | 0 | 74
  4 | 0 | 0 | 35 | 35
  4.5 | 58 | 48 | 0 | 106
  5 | 0 | 0 | 7 | 7
  Missing Data | 0 | 0 | 1 | 1
Procedure Type [Number; unit: participants]
  Orthopedic | 72 | 70 | 35 | 177
  General Surgery | 7 | 10 | 6 | 23
  Other | 11 | 10 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Airway Seal Pressure After Device Placement
Description: Airway seal pressure is defined as the pressure in cmH2O at which the needle of a manometer attached to the anesthesia circuit reaches equilibration, associated with an audible air leak from the subject's oropharynx or gastric insufflation, limited to a maximum pressure of 40 cmH2O. It is measured with the subject's head and neck in neutral position, the expiratory valve on the anesthesia machine closed, and the fresh gas flow set to five liters per minute.
Time Frame: Measured within 5 minutes after device placement/study initiation
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
cmH2O | 28 (6) | 27 (8) | 24 (8)

2. Secondary Outcome: Device Placement Time
Description: Device placement time is the time measured in seconds from when the study investigator picks up the airway device to confirmation of ventilation by the presence of an adequate end-tidal carbon dioxide tracing on the monitor.
Time Frame: Measured at device placement/study initiation
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
seconds | 25 (11) | 19 (9) | 21 (13)

3. Secondary Outcome: Device Placement Success Rate
Description: Device placement success rate is defined as the proportion of devices successfully placed within three attempts at device placement.
Time Frame: Measured at the time of attempted study device placement immediately after the induction of general anesthesia
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants
  Attempt 1 | 83 | 84 | 41
  Attempt 2 | 6 | 3 | 4
  Attempt 3 | 1 | 3 | 0

4. Secondary Outcome: Device Ease of Insertion
Description: Device ease of insertion is graded as either easy, slightly difficult, difficult, or impossible. The outcome measure is the proportion of successful study device placements recorded as easy versus slightly difficult versus difficult versus impossible.
Time Frame: Reported by the device operator at the time successful device placement is recorded.
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants
  Easy | 73 | 77 | 38
  Slight Difficulty | 16 | 11 | 7
  Moderate Difficulty | 0 | 0 | 0
  Difficult | 1 | 1 | 0
  Missing Data | 0 | 1 | 0

5. Secondary Outcome: Device Position in Relation to the Vocal Cords
Description: Device position in relation to the vocal cords is assessed with a flexible fiberoptic camera and graded as follows: 1 = full view of the vocal cords, 2 = partial view of the vocal cords including the arytenoids, 3 = view of the epiglottis only, and 4 = other (device cuff, pharynx or other structures).
Time Frame: Measured within 5 minutes of successful study device placement
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants
  1 | 62 | 71 | 28
  2 | 6 | 4 | 10
  3 | 14 | 7 | 4
  4 | 8 | 8 | 3

6. Secondary Outcome: Device Use Time (Min)
Description: Device Use Time is the time recorded to the nearest minute of the period bounded by the time the device placement was determined to be adequate in the study subject to its withdrawal from the study subject.
Time Frame: Measured between successful device placement and device removal for any reason, approximately 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Air-Q SP | Air-Q | I-gel
Number analyzed (Participants) | 90 | 90 | 45
minutes | 60 (34) | 65 (40) | 70 (41)

7. Secondary Outcome: Incidence of Gastric Insufflation
Description: Gastric insufflation is present when audible air sounds are heard by stethoscope over the subject's epigastrium.
Time Frame: Measured within 5 minutes of device placement/study initiation
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants | 0 | 0 | 0

8. Secondary Outcome: Incidence of Gastric Aspiration
Description: Gastric aspiration is present when gross gastric contents or bile is observed on or within the device or within the subject's oropharynx. The outcome is the proportion of study subjects in whom the outcome measure was observed.
Time Frame: Measured between successful device placement and device removal for any reason.
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants | 0 | 0 | 0

9. Secondary Outcome: Incidence of Oropharyngeal Injury
Description: Oropharyngeal injury is defined as a new lip, tongue, buccal, or pharyngeal abrasion or laceration or dental damage observed in the immediate recovery area after use of a study device.
Time Frame: Measured in the post-anesthesia care unit/recovery room within 15 minutes after device removal
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants | 2 | 0 | 1

10. Secondary Outcome: Overall Clinical Usefulness
Description: Excellent, good, fair, or inadequate. Scale defined by clinical measures and observations.
Time Frame: Reported by the device operator at the time of device removal
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants
  Excellent | 56 | 65 | 24
  Good | 6 | 4 | 1
  Fair | 27 | 21 | 20
  Inadequate | 1 | 0 | 0

11. Secondary Outcome: Oropharyngolaryngeal Morbidity at Discharge
Description: Perioperative oropharyngolaryngeal morbidity is assessed by the subject's response to standardized questions regarding oropharyngeal complaints.
Time Frame: Measured prior to discharge from phase II of the post-anesthesia care unit/recovery room
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 90 | 90 | 45
participants
  Sore Throat | 38 | 28 | 7
  Pain on Swallowing | 29 | 20 | 3
  Pain in Jaw | 1 | 0 | 0
  Pain in Mouth | 2 | 1 | 0
  Pain on Speaking | 2 | 3 | 0
  Tongue Swelling | 2 | 2 | 1
  Tongue Numbness | 2 | 2 | 1
  Face Numbness | 2 | 2 | 0
  Lip Numbness | 4 | 3 | 1
  Ear Pain | 2 | 4 | 0
  Hearing Change | 1 | 0 | 0

12. Secondary Outcome: Oropharyngolaryngeal Morbidity at 24 Hours Post-operatively
Description: as for outcome 11
Time Frame: Measured at 24 hours after device placement/study initiation
Measure: Number; unit: participants
Arm/Group | Air-Q | Air-Q SP | I-gel
Number analyzed (Participants) | 86 | 87 | 43
participants
  Sore Throat | 42 | 50 | 15
  Pain on Swallowing | 37 | 37 | 7
  Pain in Jaw | 3 | 2 | 2
  Pain in Mouth | 6 | 1 | 1
  Pain on Speaking | 4 | 2 | 2
  Tongue Swelling | 1 | 1 | 0
  Tongue Numbness | 1 | 0 | 3
  Face Numbness | 0 | 0 | 0
  Lip Numbness | 4 | 2 | 1
  Ear Pain | 1 | 2 | 1
  Hearing Change | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Up to 24 hours post-device use
Description: Note: "Other" adverse events include any subject experiencing any non-serious adverse event not included as a secondary outcome measure on post-procedure questioning at any time point up to 24 hours post-device use.
Arm/Group | Air-Q | Air-Q SP | I-gel
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/45
Other Adverse Events (participants affected / at risk) | 1/90 | 1/90 | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Air-Q (N=90) | Air-Q SP (N=90) | I-gel (N=45)
Lip swelling/bruise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Any reported or observed swelling or bruise of either the upper or lower lip.
Oropharyngeal bruise (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Any reported or observed bruise within the oral cavity or posterior pharynx
Oropharyngeal heme/blood (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Any reported or observed blood, including trace amounts, in the oral cavity or posterior pharynx.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No